CLINICAL TRIAL: NCT06646393
Title: The Effect of Paternal Skin-to-Skin Contact on Breastfeeding Process After Cesarean Section:A Randomized Controlled Trial
Brief Title: The Effect of Paternal Skin-to-Skin Contact on Breastfeeding Process After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Emine Serap ÇAĞAN, Principal Investigator, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AgriIbrahimCec
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2023-04

CONDITIONS: Skin to Skin Contact; Skin to Skin Contact in Cesarean Deliveries
Keywords: skin to skin contact; paternal; breastfeeding; cesarean section
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Father-baby skin-to-skin contact was applied within the first hour immediately after the cesarean delivery. During the Father-Baby Skin-to-Skin Contact stage, the newborns were laid face down on their father's bare chest and covered with a blanket.
Who Masked: Outcomes Assessor
Masking Description: The skin-to-skin group received skin-to-skin contact from a midwife working in the clinic. The outcome assessor is not aware of the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paternal skin to skin contact group (Experimental): Father-baby skin-to-skin contact was applied within the first hour immediately after the cesarean delivery. During the Father-Baby Skin-to-Skin Contact stage, the newborns were laid face down on their father's bare chest and covered with a blanket.
  Interventions: Other: Skin to skin contact
- Control group (No Intervention): Routine care was given to the control group. After the mothers' procedures were completed, the breastfeeding process was started.

INTERVENTIONS:
Other: Skin to skin contact — Father-baby skin-to-skin contact was applied within the first hour immediately after the cesarean delivery. During the Father-Baby Skin-to-Skin Contact stage, the newborns were laid face down on their father's bare chest and covered with a blanket.
  Arms: Paternal skin to skin contact group

SUMMARY:
This study aims to investigate the effect of paternal skin contact on breastfeeding after cesarean section.The research was conducted at Ağrı Training and Research Hospital, Gynecology and Obstetrics Clinic between April 2023 and August 2023.A total of 126 mothers who gave birth by cesarean section, their spouses and newborns, 61 in the skin-to-skin contact group and 65 in the control group, participated in the study. Randomization of the groups participating in the study was done by simple random method using the website www.random.org.The socio-demographic characteristics introduction form, the questionnaire regarding skin-to-skin contact and breastfeeding process, and the LATCH Breastfeeding and Diagnostic Measurement Tool were used to collect research data.

DETAILED DESCRIPTION:
The research was conducted in two groups: skin contact group and control group. This study aims to investigate the effect of paternal skin contact on breastfeeding after cesarean section.The research was conducted at Ağrı Training and Research Hospital, Gynecology and Obstetrics Clinic between April 2023 and August 2023.A total of 126 mothers who gave birth by cesarean section, their spouses and newborns, 61 in the skin-to-skin contact group and 65 in the control group, participated in the study. Randomization of the groups participating in the study was done by simple random method using the website www.random.org.The socio-demographic characteristics introduction form, the questionnaire regarding skin-to-skin contact and breastfeeding process, and the LATCH Breastfeeding and Diagnostic Measurement Tool were used to collect research data.

ELIGIBILITY:
Inclusion Criteria:

* Caesarean section
* single and live birth
* giving birth between 38-40 weeks
* not having a mental or physical barrier to breastfeeding,
* not having a need for neonatal intensive care in the baby,
* not having a condition that prevents breastfeeding in the baby,
* not having a condition that prevents skin contact with the baby
* agreeing to participate in the research

Exclusion Criteria:

* Having a vaginal birth
* Having a premature birth
* Having a mental or physical disability that prevents breastfeeding
* Having the baby referred to neonatal intensive care
* Having a condition that prevents breastfeeding
* Having a condition that prevents skin-to-skin contact

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
LATCH breastfeeding diagnostic scale | after skin contact and before discharge
  by observing breastfeeding; It is an assessment tool that is quick and easy to apply, created to detect problems that may occur during breastfeeding. Scoring is done between 0-2 and the maximum score that can be obtained is 10. In the non-breakpoint measurement tool, a high score indicates successful breastfeeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Agri Ibrahim Cecen University, Ağrı, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided